CLINICAL TRIAL: NCT00733785
Title: An Open-Label, Randomized, Crossover Study to the Dose Proportionality of RSG XR in Healthy Volunteers in Fasting Conditions
Brief Title: PK, Dose Proportionality, Food Effect And Repeat Dose Study Of Rosiglitazone XR In Healthy Volunteers
Acronym: Rosi XR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AVA109939
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
Keywords: Rosiglitazone XR; Pharmacokinetics; Strength Equivalence.; Alzheimers Disease; Repeat dose; Dose proportionality
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 2mg tablet (Experimental): 2 mg tablet fasted
  Interventions: Drug: Rosiglitazone XR
- 4 mg tablet (Experimental): 4 mg tablet fasted
  Interventions: Drug: Rosiglitazone XR
- 8mg tablet (Experimental): 8 mg tablet fasted
  Interventions: Drug: Rosiglitazone XR
- 2 x 4 mg tablets (Experimental): 2 x 4mg tablets fasting
  Interventions: Drug: Rosiglitazone XR
- 2 x 2mg tablets (Experimental): 2 x 2mg tablets fasting
  Interventions: Drug: Rosiglitazone XR
- 8 mg tablet fed (Experimental): 8 mg tablet fed
  Interventions: Drug: Rosiglitazone XR
- Repeat dose (Experimental): 8 mg once a day for 6 days
  Interventions: Drug: Rosiglitazone XR

INTERVENTIONS:
Drug: Rosiglitazone XR — Rosiglitazone extended release formulation

SUMMARY:
The present pharmacokinetic study is designed to further characterise the pharmacokinetics of the RSG XR formulation and aims to assess dose proportionality, strength equivalence, the food effect and the pharmacokinetics after repeat dosing.

DETAILED DESCRIPTION:
The present pharmacokinetic study is designed to further characterise the pharmacokinetics of the RSG XR formulation manufactured in Crawley and aims to assess dose proportionality, strength equivalence, the food effect and the pharmacokinetics after repeat dosing. The study aims to enroll sufficient number of subjects to ensure 48 subjects complete Study Part 1 (6 period crossover design) and a further 12 subjects complete Study Part 2 (repeat dosing).

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

Healthy male and female (not gender stratified) subjects aged 18-55 years inclusive - healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, ECGs, and other tests. A subject with clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator and the GSK Medical Monitor considers that the findings will not introduce additional risk factors and will not interfere with the study procedures.

Body weight greater than 50 kg (110lbs and Body mass index (BMI) between 19 and 30 kg/m2 Willing and able to give written informed consent, willing to participate for the full duration of the study, and able to understand and follow instructions related to study procedures.

Female subjects able to bear children must agree to use an adequate method of contraception for the duration of the study and for 14 days after last dose (see for details of highly effective methods to avoid pregnancy). Female subjects who are pre-menopausal or who have been post-menopausal for less than 2 years must undertake pregnancy testing (serum test) less than or equal to 7 days before Visit 1, which must be negative

Females, who are on hormone replacement therapy (HRT), and whose menopausal status is in doubt, will be required to use a highly effective method to avoid pregnancy, as outlined in the protocol, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a highly effective method to avoid pregnancy.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Any clinically relevant abnormality identified on the screening history and physical or laboratory examination or any other medical condition or circumstance making the volunteer unsuitable for participation in the study. Specific examples include, coronary artery disease, myocardial infarction, congestive heart failure, type 2 diabetes, renal disease and hypertension. If there is doubt on the appropriateness of a subject, that subject's eligibility for the study must be reviewed with the medical monitor prior to enrolment.

History of surgical procedures that might affect the absorption of rosiglitazone (e.g., partial/total gastrectomy, cholecystectomy) or any hepatic or biliary abnormalities such as Gilbert's syndrome.

History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 150mls of wine or 360mls of beer or 45mls of hard liquor) within 6 months of screening.

Subject smoking more than 10 cigarettes per day. Positive urine drug screen (UDS) including alcohol at screening or check-in visits.

Positive hepatitis B virus, hepatitis C virus or HIV test at screening. Positive serum beta-human chorionic gonadotropin test (females). Women who are pregnant, lactating, or planning to become pregnant. Male subjects who are not willing to abstain from or use a condom during sexual intercourse with pregnant or lactating females. Male subjects not willing to use a condom, plus another form of contraception (e.g., spermicide, IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a female who could become pregnant. Male subjects not willing to adhere to these contraceptive criteria from administration of study medication until completion of follow-up procedures.

Female subjects not willing to use proposed contraceptive methods. Use of prescription or non-prescription drugs [in particular known inhibitors of cytochrome 2C8 (Gemfibrozil, trimethoprim, glitazone, monteleucast, quercetin) or inducer (rifampin)], vitamins, herbal and dietary supplements (including St. John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Excluded from this list are acetaminophen and paracetamol at doses of less than or equal to 2 grams/day, thyroid replacement therapy, and hormonal methods of contraception (including oral contraceptives, injectable progesterone, progestin subdermal implants and progesterone-releasing IUDs, but NOT postcoital contraceptive methods) and hormone replacement therapy which will be permitted throughout the study.

Donation of blood in excess of 500 mL within 56 days prior to first dose of study medication.

History of sensitivity to heparin, heparin-induced thrombocytopenia or sensitivity to any of the study medications or components thereof.

History of hypersensitivity to rosiglitazone, or any of the excipients in the formulations.

Systolic BP greater than 140 mm Hg and/or Diastolic BP greater than 90 mm Hg at screening or check-in.

QTc (machine read) greater than 450 ms on the screening ECG. History of glucose intolerance (serum glucose greater than 110 mg/dl or 6.1 mmol/L after 8 hours fasting) Subjects have had treatment with a new molecular entity (investigational drug) or any other trial during the previous 30 days or five half-lives, whichever is longer. (the washout is from last dose of study medication in the previous study until the first dose of study medication).

Current evidence of drug abuse or history of drug abuse within one year of allocation Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.

Vulnerable subjects (e.g. persons kept in detention).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08-13 (Actual); Primary Completion 2008-11-28 (Actual); Study Completion 2008-11-28 (Actual)

PRIMARY OUTCOMES:
•For the single dose period: AUC(0-inf) and Cmax of RSG XR.•For repeat dose period on Day 1 and 6:, AUC(0-24) and Cmax of RSG XR. | Single dose and Day 6 for repeat dose

SECONDARY OUTCOMES:
For single dose period: AUC(0-t), Tmax, lz, and t1/2 of RSG XR as data permit | Single dose and Day 6 for repeat dose
For repeat dose period: Tmax, concentration at the end of the dosing interval (Ct), minimum observed concentration (Cmin), | 6 days
Average concentration during a dosing interval (Cav), t1/2, , accumulation ratio(Rs) Rs= (AUC(0-t) last day)/(AUC(0-t) first day) and degree of fluctuation DF= (Cmax-Cmin)/Cave. | 6 days
• Safety reporting (adverse events, laboratory testing, ECG, vital signs) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study AVA109939 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/AVA109939?search=study&search_terms=AVA109939#rs